CLINICAL TRIAL: NCT00562861
Title: Treatment for Bipolar Depression: Acute & Prophylactic Efficacy With Citalopram
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MH78060-01A1; 5R01MH078060-04 (NIH)
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Results first posted 2017-02-13 (Actual); Last update posted 2017-03-24 (Actual); Status verified 2017-02

CONDITIONS: Bipolar Disorder; Bipolar Depression
Keywords: Bipolar Disorder; Bipolar Depression; Clinical Trials, Phase II; Clinical Pharmacology
MeSH Terms: conditions — Bipolar Disorder | interventions — Citalopram; Lithium; Lamotrigine; Valproic Acid; Carbamazepine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- citalopram + mood stabilizer (Active Comparator): All patients are on baseline mood stabilizers and are randomized to receive citalopram or placebo. In this arm, they are randomly assigned to citalopram.
  Interventions: Drug: citalopram + mood stabilizer
- placebo + mood stabilizer (Placebo Comparator): All patients are on baseline mood stabilizers and are randomized to receive citalopram or placebo. In this arm, they are randomly assigned to placebo
  Interventions: Drug: placebo + mood stabilizer

INTERVENTIONS:
Drug: citalopram + mood stabilizer — Citalopram dose will be flexibly designed, beginning at 10 mg/d for at least one week, and the increased by 10 mg per week to a maximum of 50 mg/d. No target dose will be provided but rather clinicians will dose to clinical efficacy. Thus the study will provide clinicians data on the effective dose if it is positive. The dose will not be predetermined at static amounts.
  Other Names: Celexa
  Arms: citalopram + mood stabilizer
Drug: placebo + mood stabilizer — This arm will only receive mood stabilizing medication. All subjects will be required to receive treatment with lithium, lamotrigine, valproate, or carbamazepine for at least one month at therapeutic blood levels or doses before randomization, or they must initiate one of these agents at study entry.
  Other Names: lithium, lamotrigine, valproate, or carbamazepine
  Arms: placebo + mood stabilizer

SUMMARY:
Bipolar depression is one of the least studied depressive illnesses. The standard practice for many doctors is to use antidepressant medicines, but there are few studies on the long-term results of these medicines. The goal of this study is to look at how effective and safe these medicines are in treating bipolar depression when taken with a mood stabilizer medicine.

The drug being studied is citalopram, also known as Celexa. Celexa is FDA approved for the treatment of major depression, but is not FDA approved for the treatment of bipolar depression. It is, however, standard practice for many doctors is to use antidepressants, like Celexa, to treat their patients with bipolar disorder depression.

The drug will be studied in three ways. We will see if it helps treat depressive symptoms. We will see how the drug affects the brain using PET and fMRI scans. Finally, we will look at the possibility that there may be a gene that could predict if a person would get better taking the drug using genetics.

DETAILED DESCRIPTION:
The problem of interest

Depression is a common serious illness, with great personal suffering and a 10% or more risk of suicide. There are two kinds of depression, bipolar (depression alternating with mood swings) and unipolar ("simple" depression, or major depressive disorder). In both kinds of depression, antidepressants are commonly used. However, unlike unipolar depression, where a good deal of research supports this use, there is very little research on antidepressant use in bipolar disorder. Some studies support benefit with antidepressants for bipolar depression; i.e., if one is depressed, antidepressants can help a patient get better in the short-term. However, long-term studies are limited; the few available studies with older antidepressants did not demonstrate long-term preventive benefit. Some clinicians think new generation antidepressants (like Prozac and other serotonin reuptake inhibitors) are safer and more effective than the older antidepressants. Yet there are no rigorous long-term studies of new generation antidepressants in bipolar disorder. Recent observational studies with new antidepressants suggest that they may be harmful to some patients with bipolar disorder.

Clinicians are thus left in a quandary. Antidepressants appear to be effective in the short term, but should the antidepressants (especially new generation antidepressants) be continued long-term? Some studies support both approaches. Importantly, some evidence exists that antidepressants can make many patients worse, with more and more depression or mania over time.

This is a major public health problem, since clinicians prescribe antidepressants for the long-term in up to 80% of patients with bipolar disorder. This represents standard treatment, despite the limitations of the available evidence and the suggestion that in some patients such antidepressant use may be harmful.

This study is also looking at possible biological predictors that may reflect an individual patients' likelihood that he or she will respond to a specific treatment.

How the problem will be studied

This project is one of the most rigorous studies of new generation antidepressants in long-term treatment of bipolar disorder. We will recruit patients with bipolar disorder who are currently in a depressive episode and are taking or eligible and interested in taking a mood stabilizer such as lithium. Subjects will then be randomly put into one of two groups. The first group will receive the generic antidepressant, citalopram while the other group will receive placebo, sugar pill. Patients will be closely followed and monitored by the research psychiatrist and through a series of safety labs. Subjects will have an MRI and PET scan for the biological predictors section of the study. The key question is: After the acute recovery, should they continue antidepressants or not?

As there is limited scientific data, and opposing kinds of clinical experience, there is no clear rationale to making this decision. Our study seeks to provide a scientific basis for making that decision. We plan to follow subjects for a goal of 1 year to obtain long-term outcome data on which approach is best.

How the research will advance scientific knowledge or human health

Since there are no rigorous long-term studies with new generation antidepressants in bipolar disorder, this study will be a major advance in that knowledge. Clinicians will have some evidence on which to base that decision, rather than simply their own opinions or patients' preferences. In the light of recent evidence that antidepressants are potentially harmful to some patients, this study will provide more information about how new antidepressants work specifically for bipolar patients rather than unipolar depression (also known as major depression). The biological portion of the study will shed light on possible biological factors that could show how an individual may respond to a specific treatment. This could potentially help doctors to decide on which treatments are more or less likely to work for their individual patients rather then using a "hit or miss" type method.

ELIGIBILITY:
Inclusion Criteria:

* Current age ≥18 years
* DSM-IV diagnosis of BPD, type-I, or type-II
* Current major depressive episode using DSM-IV criteria, lasting 8 weeks or longer.
* Use of lithium, divalproex, carbamazepine, or lamotrigine at therapeutic serum levels or doses for ≥4 weeks prior to study entry, or willingness to accept one of these agents.
* Prior to initial evaluations, each subject must provide competent, written, informed consent.

Exclusion Criteria:

* Past non-response to a therapeutic trial of R,S-citalopram (≥100 mg/day for ≥8 weeks).
* Previous intolerance of R,S-citalopram;
* Diagnosis of unipolar depression
* Diagnosis of schizoaffective disorder
* Serious medical illness with acute instability (cardiac, respiratory, hepatic, renal), based on hospitalization in the past month
* Abnormal thyroid function tests
* Previous allergic reaction to or inability to tolerate lithium, divalproex, or carbamazepine at therapeutic serum levels.
* Current or past renal dysfunction if taking lithium
* Current or past hepatitis or other liver disease if taking divalproex
* Current or past hematologic disease if on carbamazepine
* Severe suicidal ideation, plan or intent, as documented by a score of ≥4 on the Montgomery Åsberg Depression Rating Scale suicidality item (Item 10).
* Presence of psychosis
* Cognitive impairment sufficient to impair ability to give informed consent.
* Current pregnancy, or inability to utilize contraception
* The presence of any metallic implants
* History of claustrophobia

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2007-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassir Ghaemi, MD, MPH, Principal Investigator — Tufts University Medical
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghaemi SN, Whitham EA, Vohringer PA, Barroilhet SA, Amerio A, Sverdlov O, Patkar AA. Citalopram for Acute and Preventive Efficacy in Bipolar Depression (CAPE-BD): A Randomized, Double-Blind, Placebo-Controlled Trial. J Clin Psychiatry. 2021 Jan 12;82(1):19m13136. doi: 10.4088/JCP.19m13136. PMID 33434956

RESULTS

PARTICIPANT FLOW:
Groups:
- Mood Stabilizer Plus Citalopram: citalopram + mood stabilizer: Citalopram dose will be flexibly designed, beginning at 10 mg/d for at least one week, and the increased by 10 mg per week to a maximum of 50 mg/d.
- Mood Stabilizer Plus Placebo: Mood stabilizer alone will be the treatment, with placebo used instead of double-blind citalopram.
Period: Overall Study
Arm/Group | Mood Stabilizer Plus Citalopram | Mood Stabilizer Plus Placebo
Started | 60 | 59
Completed | 40 | 48
Not Completed | 20 | 11
Not completed — Adverse Event | 1 | 1
Not completed — Lack of Efficacy | 5 | 5
Not completed — noncompliance, moved | 7 | 2
Not completed — Lost to Follow-up | 7 | 3

BASELINE CHARACTERISTICS:
Population: These subjects met inclusion/exclusion criteria and were randomized to citalopram versus placebo.
Groups:
- Mood Stabilizer Plus Citalopram: citalopram + mood stabilizer: Subjects receive the active drug, added to standard mood stabilizers.
- Mood Stabilizer Plus Placebo: Placebo plus mood stabilizer: subjects receive placebo, added to standard mood stabilizers
- Total: Total of all reporting groups
Arm/Group | Mood Stabilizer Plus Citalopram | Mood Stabilizer Plus Placebo | Total
Number analyzed (Participants) | 60 | 59 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.9 (12.6) | 42.1 (11.3) | 41.5 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 31 | 74
  Male | 17 | 28 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 21 | 20 | 41
  White | 36 | 35 | 71
  More than one race | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 60 | 59 | 119

OUTCOME MEASURES:

1. Primary Outcome: MADRS Rating Scale Change
Description: Montgomery Asberg Depression Rating scale assessed in mixed effects regression model. The total range for the scale is 0 to 60. Lower values involve less depression, while higher values involve worse depression. The change in the MADRS scale is interpreted as higher values meaning better outcomes, because more depressive symptoms are improved.
Time Frame: 6 weeks
Population: All patients randomized were analyzed in intent to treat manner.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Citalopram: Mood stabilizers given as part of standard treatment plus double-blind citalopram
- Placebo: Mood stabilizers given as part of standard treatment plus double-blind placebo
Arm/Group | Citalopram | Placebo
Number analyzed (Participants) | 60 | 59
units on a scale | 13.1 (8.4) | 15.2 (9.9)
Statistical Analysis 1: Comparison: Citalopram vs Placebo; Test type: Superiority or Other; p = 0.17, Mixed Models Analysis; F value = 1.88

ADVERSE EVENTS:
Time Frame: Adverse events are reported for 1 year of follow-up during the randomized trial.
Description: All patients were systematically interviewed for the adverse events reported.
Arm/Group | Citalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/59
Other Adverse Events (participants affected / at risk) | 23/60 | 15/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=60) | Placebo (N=59)
suicide (Psychiatric disorders) | 1 (1) | 0 (0) — Subject committed suicide which was judged to be unrelated to administration of citalopram after review by investigators and evaluation by institutional review board.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Citalopram (N=60) | Placebo (N=59)
sedation (Psychiatric disorders) | 8 (8) | 3 (3)
dry mouth (Nervous system disorders) | 6 (6) | 0 (0)
sexual dysfunction (Nervous system disorders) | 5 (5) | 0 (0)
headache (Nervous system disorders) | 4 (4) | 6 (6)
nausea (Gastrointestinal disorders) | 3 (3) | 6 (6)
diarrhea (Gastrointestinal disorders) | 1 (1) | 5 (5)
tremor (Nervous system disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No